CLINICAL TRIAL: NCT06939127
Title: A Prospective Phase II Study to Explore the Efficacy and Safety of Cryoablation Combined With Tislelizumab and Chemotherapy as Neoadjuvant Treatment, Followed by Adjuvant Tislelizumab Therapy in Resectable Stage II-IIIB Non-small Cell Lung Cancer
Brief Title: Cryoablation Combined With Tislelizumab and Chemotherapy as Neoadjuvant and Adjuvant Therapy in Resectable Stage II-IIIB NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Dongsheng Yue, Chief Physician of Surgery, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONCEPT study
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
Keywords: II-III NSCLC; neoadjuvant; adjuvant; pathological complete response
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Drug Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cryoablation Combined with Tislelizumab (Experimental): Neoadjuvant Phase:
  Eligible patients first undergo cryoablation of the primary tumor. Then, 7±3 days after cryoablation, they start treatment with tislelizumab (200 mg) plus platinum-based doublet chemotherapy, given every 3 weeks for 3-4 cycles.
  Surgery should be performed as soon as possible within 4-6 weeks after the last dose of neoadjuvant therapy.
  Adjuvant Phase:
  The first dose of tislelizumab (cycle 1 of the adjuvant phase) should be administered within 2-8 weeks after surgery. Patients will continue to receive tislelizumab (400 mg, Q6W) as adjuvant therapy every 6 weeks until one of the following events occurs: completion of 8 cycles of tislelizumab adjuvant therapy, disease recurrence, unacceptable adverse events (AEs), death, or decision by the patient and/or investigator to discontinue study treatment.
  Interventions: Drug: Neoadjuvant Cryoablation Combined with Tislelizumab and Chemotherapy; Procedure: Surgery; Drug: Adjuvant tislelizumab

INTERVENTIONS:
Drug: Neoadjuvant Cryoablation Combined with Tislelizumab and Chemotherapy — Eligible patients will start the study treatment (7-14 days between pathological diagnosis and cryoablation). Patients first undergo cryoablation of the primary tumor. Then, 7±3 days after cryoablation, they start treatment with tislelizumab (200 mg) plus platinum-based doublet chemotherapy, given every 3 weeks for 3-4 cycles.
  The following platinum-based doublet chemotherapy regimens are allowed in this trial:
  * Cisplatin/carboplatin + pemetrexed (non-squamous NSCLC)
  * Cisplatin/carboplatin + albumin-bound paclitaxel/paclitaxel (squamous NSCLC)
Procedure: Surgery — After completing neoadjuvant therapy, surgery should be performed as soon as possible within 4-6 weeks after the last dose of neoadjuvant therapy.
Drug: Adjuvant tislelizumab — Patients receiving adjuvant therapy must meet the following criteria:
  * ECOG performance status score of 0 or 1
  * Recovery from surgery and adequate organ function as determined by the investigator based on laboratory values During the adjuvant phase, patients will receive tislelizumab as adjuvant therapy. The first dose of tislelizumab (cycle 1 of the adjuvant phase) should be administered within 2-8 weeks after surgery. Patients will continue to receive tislelizumab (400 mg, Q6W) as adjuvant therapy every 6 weeks until one of the following events occurs: completion of 8 cycles of tislelizumab adjuvant therapy, disease recurrence, unacceptable adverse events (AEs), death, or decision by the patient and/or investigator to discontinue study treatment.

SUMMARY:
This is a Phase II single-arm study designed to evaluate the efficacy and safety of cryoablation combined with tislelizumab and platinum-based doublet chemotherapy as neoadjuvant therapy, followed by adjuvant tislelizumab therapy in patients with resectable stage II-IIIB non-small cell lung cancer (NSCLC).

The study consists of a screening phase, a treatment phase (including the neoadjuvant stage, surgery, and adjuvant stage), a safety follow-up period, and a survival follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at informed consent signing.
* ECOG performance status of 0 or 1.
* Histologically confirmed stage II-IIIB NSCLC (AJCC 9th edition).
* Tumor size ≤5 cm.
* Deemed suitable for R0 resection by a thoracic surgeon for radical treatment.
* Adequate cardiopulmonary function for radical surgical resection.
* Eligible for cryoablation and platinum-based doublet chemotherapy.
* Adequate blood and organ function, as per laboratory tests within 14 days before enrollment.

Exclusion Criteria:

* Prior treatment for current lung cancer, including chemotherapy or radiotherapy.
* LCNEC diagnosis.
* Known EGFR mutations or ALK translocations. For non-squamous NSCLC, EGFR mutation status must be confirmed locally or centrally if unknown.

For squamous NSCLC, EGFR testing is not required if status is unknown. ALK translocation testing is not required if status is unknown.

* Locally advanced, unresectable disease, regardless of stage or metastasis (stage IV). Patients with mediastinal lymph node involvement on CT must undergo sampling for clinical staging to exclude stage IIIB/C.
* History of interstitial lung disease, non-infectious pneumonitis, or uncontrolled pulmonary fibrosis.
* Severe chronic or active infections requiring systemic antimicrobials, including tuberculosis.
* Hospitalization for severe infections within 4 weeks before enrollment. Systemic antibiotic treatment within 2 weeks before enrollment.
* Active autoimmune disease or history of recurrent autoimmune disease.
* Exceptions: Well-controlled type 1 diabetes, hypothyroidism on hormone replacement, celiac disease, skin conditions not requiring systemic therapy, or diseases unlikely to recur without provocation.
* Severe infections requiring systemic treatment within the past 4 weeks.
* Corticosteroid or immunosuppressive use within 14 days before enrollment, except for specific local, topical, or short-term uses.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | Up to approximately 8 weeks following completion of neoadjuvant treatment
  pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to Study Week 15 (before surgery)
  ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1 before surgery.
Radiological downstaging rate | Up to Study Week 15 (before surgery)
  The proportion of patients with radiological T, N, and overall stage reduction (AJCC v9) compared to baseline after neoadjuvant therapy.
Major Pathological Response (mPR) Rate | Up to approximately 8 weeks following completion of neoadjuvant treatment
  mPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy.
Event Free Survival (EFS) | Up to approximately 2 years
  EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause. EFS determined either by biopsy assessed by local pathologist or by investigator-assessed imaging using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Overall Survival (OS) | Up to approximately 2 years
  OS is defined as the time from randomization until death from any cause.
Number of participants experiencing treatment-emergent adverse events (TEAEs) | Up to approximately 2 years
  An AE was defined as any untoward medical occurrence in a study participant administered study drug and which does not necessarily have to have a causal relationship with this study drug. The number of participants who experienced an AE is presented.
Change From Baseline in Neoadjuvant and Adjuvant Phase in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Baseline, during the neoadjuvant phase (Cycle 3), during the adjuvant phase (Cycles 1, 3, 5, and 7), and during safety follow-up visits (up to 2 years)
  Change from baseline in QoL score using the EORTC QLQ-C30 will be determined. The EORTC QLQ-C30 is the most widely used cancer-specific, health-related QoL instrument comprised of 30 individual items arranged as both multi-item scales and individual items. Specifically, these items are divided into 5 functional scales (15 items total), 3 symptom scales (7 items total), 6 individual items.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Yue Chief Physician of Surgery, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No